CLINICAL TRIAL: NCT05541978
Title: Thrombosis in Newly Diagnosed Multiple Myeloma Patients: a Clinical Audit of Intermediate Dose Low Molecular Weight Heparin
Brief Title: Thrombosis in Patients With Multiple Myeloma in an University Medical Center
Acronym: THRIMM
Status: Completed | Type: Observational
Sponsor: Catalina Codreanu (Other)
Responsible Party: Sponsor-Investigator, Catalina Codreanu, Master student, Medicine, University Medical Center Groningen
Organization: University Medical Center Groningen (Other)
Other Study IDs: 202200311
Record Dates: First submitted 2022-09-12; First posted 2022-09-15 (Actual); Last update posted 2023-07-03 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma; Venous Thromboembolism; Arterial Thromboembolism
MeSH Terms: conditions — Multiple Myeloma; Venous Thromboembolism

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Multiple myeloma — We will explore the multiple myeloma associated thrombosis risk.

SUMMARY:
Main research question:

What is the present venous thrombosis incidence and what are the current practices of prescribing thromboprophylaxis in patients with multiple myeloma (MM)?

Design:

The present study is a retrospective cohort study. The patients will be selected from the electronic patient dossier (EPD) of the University Medical Center Groningen (UMCG). The present study will include newly diagnosed adult patients with a first MM at the UMCG between 1st of January 2014 and 1st of September 2021. The primary outcome of the study is the incidence of venous thromboembolism (VTE) with one year of diagnosis of MM. The investigators will also describe the various thromboprophylaxis regimens used and their corresponding VTE incidence. The secondary outcome will be the incidence of arterial thrombosis (AT) within the same period of time. Possible confounders are the therapy administered for MM, thromboprophylaxis type, age and patient comorbidities. Lastly, the third outcome will be a description of current thromboprophylaxis practices in the UMCG. Each outcome will be described separately.

Expected results:

Based on the study by de Waal et al in which they included 474 MM patients treated at the UMCG and at 4 hospitals in the province Friesland, the investigators expect to record a VTE incidence of approximately 15%.

DETAILED DESCRIPTION:
Background:

Multiple myeloma (MM) is a neoplastic clonal proliferation of plasma cells causing a considerable worldwide burden of disease. In 2016 Western Europe was one of the regions with the highest MM incidence globally, with an age-standardized incidence of 4.6 per 100.000 (95% UI, 3.7-5.5). MM is associated with multiple complications which make the management of this disease particularly difficult. Moreover, patients with MM have a raised risk of venous thromboembolism (VTE) which substantially increases their mortality risk. The link between malignancy and the development of a hypercoagulable state has been extensively studied, with altered coagulation, patient comorbidities, tumour characteristics and treatment side-effects all playing a role in the pathogenesis of thrombosis in cancer. Specifically in MM, the increased VTE risk seems to be partially due to aberrations in haemostasis, such as acquired activated Protein C resistance and increased levels of Factor VIII and Von Willebrand Factor.

MM treatment and maintenance therapy has developed and improved substantially during the past decades, with immunomodulatory drugs (IMIDs), namely lenalidomide- or thalidomide-based regimens, being currently the most effective and used option. Nevertheless, one of the challenges of these regimens remains the associated elevated VTE risk, which is especially high in newly diagnosed MM patients treated with IMIDs and dexamethasone. Various mechanisms have been researched to explain the increased VTE risk. For instance, transiently decreased thrombomodulin levels during the first months of treatment have been associated with an increased thrombosis risk during the initial period of therapy. Moreover, high levels of cathepsin G have also been hypothesized to contribute to the high thrombosis incidence in MM patients undergoing treatment.

Choosing an appropriate thromboprophylaxis regimen in MM patients treated with IMIDs remains a challenge in clinical practice. Randomized controlled trials (RCTs) did not show a difference in the VTE risk between the use of aspirin or low molecular weight heparin (LMWH) in the management of MM patients. Furthermore, despite thromboprophylaxis, high VTE incidence remains a concerning problem in contemporary lenalidomide-based regimens. Therefore, the current study seeks to describe the use and efficacy of current thromboprophlaxis regimens in MM patients treated with IMIDs in an university medical center in order to assess the current VTE incidence and the effectiveness of thromboprophylaxis protocols in place.

Research question:

What is the present venous thrombosis incidence and what are the current practices of prescribing thromboprophylaxis in patients with multiple myeloma?

Design:

The present study is a retrospective cohort study. The patients will be selected from the electronic patient dossier (EPD) of the University Medical Center Groningen (UMCG). The present study will include newly diagnosed adult patients with a first MM at the UMCG between the 1st of January 2014 and 1st of September 2021. The primary outcome of the study is the incidence of VTE with one year of diagnosis of MM. The investigators will also describe the various thromboprophylaxis regimens used and their corresponding VTE incidence. The secondary outcome will be the incidence of arterial thrombosis (AT) within the same period of time. Possible confounders are the therapy administered for MM, thromboprophylaxis type, age and patient comorbidities. Lastly, the third outcome will be a description of current thromboprophylaxis practices in the UMCG. Each outcome will be described separately.

Expected results:

Based on the study by de Waal et al in which they included 474 MM patients treated at the UMCG and at 4 hospitals in the province Friesland, the investigators expect to record a VTE incidence of approximately 15%.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients diagnosed with multiple myeloma between 1st of January 2014 and 1st of September 2021
* Patients diagnosed at UMCG
* Patients diagnosed with multiple myeloma based on the IMWG criteria

Exclusion Criteria:

* Patients first diagnosed with multiple myeloma before 1st of January 2014
* Patients diagnosed after 1st of September 2021
* Patients diagnosed with a relapse of multiple myeloma between 1st of January 2014 and 1st of September 2021 of a multiple myeloma diagnosed <2014
* Patients who are marked as objecting to the use of their data for research purposes in the electronic patient dossier of UMCG

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This study seeks to include all available multiple myeloma patients treated in the UMCG. The inclusion of all patients is necessary in order to be able to calculate the incidence of venous thrombosis and in order to describe the use of thromboprophylaxis in these patients. Therefore all UCMG patients qualifying based on the inclusion and exclusion criteria will be included. We approximate that there are 60 new cases of multiple myeloma diagnosed per year in the UMCG. Thus, around 480 patients would be included in the study.
Sampling Method: Non-Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2022-09-01 (Actual); Primary Completion 2023-02-01 (Actual); Study Completion 2023-03-01 (Actual)

PRIMARY OUTCOMES:
Venous thromboembolism incidence | 1 year
  We will calculate the incidence of venous thromboembolism of patients within one year of a first diagnosis of multiple myeloma. The influence of various risk factors will be investigated.

SECONDARY OUTCOMES:
Arterial thromboembolism | 1 year
  We will calculate the incidence of arterial thromboembolism of patients within one year of a first diagnosis of multiple myeloma. The influence of various risk factors will be investigated.

OTHER OUTCOMES:
Frequency of thrombosis events per thromboprophylaxis regimen | 1 year
  We will investigate the frequency of thrombosis events per thromboprophylaxis regimen.

CONTACTS AND LOCATIONS:
Overall Officials: Karina Meijer, Principal Investigator — University Medical Center Groningen
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands

REFERENCES:
- [Background] Cowan AJ, Allen C, Barac A, Basaleem H, Bensenor I, Curado MP, Foreman K, Gupta R, Harvey J, Hosgood HD, Jakovljevic M, Khader Y, Linn S, Lad D, Mantovani L, Nong VM, Mokdad A, Naghavi M, Postma M, Roshandel G, Shackelford K, Sisay M, Nguyen CT, Tran TT, Xuan BT, Ukwaja KN, Vollset SE, Weiderpass E, Libby EN, Fitzmaurice C. Global Burden of Multiple Myeloma: A Systematic Analysis for the Global Burden of Disease Study 2016. JAMA Oncol. 2018 Sep 1;4(9):1221-1227. doi: 10.1001/jamaoncol.2018.2128. PMID 29800065
- [Background] Kristinsson SY, Pfeiffer RM, Bjorkholm M, Goldin LR, Schulman S, Blimark C, Mellqvist UH, Wahlin A, Turesson I, Landgren O. Arterial and venous thrombosis in monoclonal gammopathy of undetermined significance and multiple myeloma: a population-based study. Blood. 2010 Jun 17;115(24):4991-8. doi: 10.1182/blood-2009-11-252072. Epub 2010 Mar 18. PMID 20299513
- [Background] Schoen MW, Carson KR, Luo S, Gage BF, Li A, Afzal A, Sanfilippo KM. Venous thromboembolism in multiple myeloma is associated with increased mortality. Res Pract Thromb Haemost. 2020 Sep 25;4(7):1203-1210. doi: 10.1002/rth2.12411. eCollection 2020 Oct. PMID 33134785
- [Background] Falanga A, Donati MB. Pathogenesis of thrombosis in patients with malignancy. Int J Hematol. 2001 Feb;73(2):137-44. doi: 10.1007/BF02981929. PMID 11372723
- [Background] De Cicco M. The prothrombotic state in cancer: pathogenic mechanisms. Crit Rev Oncol Hematol. 2004 Jun;50(3):187-96. doi: 10.1016/j.critrevonc.2003.10.003. PMID 15182825
- [Background] Colombo R, Gallipoli P, Castelli R. Thrombosis and hemostatic abnormalities in hematological malignancies. Clin Lymphoma Myeloma Leuk. 2014 Dec;14(6):441-50. doi: 10.1016/j.clml.2014.05.003. Epub 2014 Jun 11. PMID 25018062
- [Background] Auwerda JJ, Sonneveld P, de Maat MP, Leebeek FW. Prothrombotic coagulation abnormalities in patients with newly diagnosed multiple myeloma. Haematologica. 2007 Feb;92(2):279-80. doi: 10.3324/haematol.10454. PMID 17296591
- [Background] Elice F, Fink L, Tricot G, Barlogie B, Zangari M. Acquired resistance to activated protein C (aAPCR) in multiple myeloma is a transitory abnormality associated with an increased risk of venous thromboembolism. Br J Haematol. 2006 Aug;134(4):399-405. doi: 10.1111/j.1365-2141.2006.06208.x. PMID 16882132
- [Background] Gay F, Jackson G, Rosinol L, Holstein SA, Moreau P, Spada S, Davies F, Lahuerta JJ, Leleu X, Bringhen S, Evangelista A, Hulin C, Panzani U, Cairns DA, Di Raimondo F, Macro M, Liberati AM, Pawlyn C, Offidani M, Spencer A, Hajek R, Terpos E, Morgan GJ, Blade J, Sonneveld P, San-Miguel J, McCarthy PL, Ludwig H, Boccadoro M, Mateos MV, Attal M. Maintenance Treatment and Survival in Patients With Myeloma: A Systematic Review and Network Meta-analysis. JAMA Oncol. 2018 Oct 1;4(10):1389-1397. doi: 10.1001/jamaoncol.2018.2961. PMID 30098165
- [Background] Carrier M, Le Gal G, Tay J, Wu C, Lee AY. Rates of venous thromboembolism in multiple myeloma patients undergoing immunomodulatory therapy with thalidomide or lenalidomide: a systematic review and meta-analysis. J Thromb Haemost. 2011 Apr;9(4):653-63. doi: 10.1111/j.1538-7836.2011.04215.x. PMID 21255254
- [Background] Qiao SK, Guo XN, Ren JH, Ren HY. Efficacy and Safety of Lenalidomide in the Treatment of Multiple Myeloma: A Systematic Review and Meta-analysis of Randomized Controlled Trials. Chin Med J (Engl). 2015 May 5;128(9):1215-22. doi: 10.4103/0366-6999.156134. PMID 25947406
- [Background] Yang B, Yu RL, Chi XH, Lu XC. Lenalidomide treatment for multiple myeloma: systematic review and meta-analysis of randomized controlled trials. PLoS One. 2013 May 14;8(5):e64354. doi: 10.1371/journal.pone.0064354. Print 2013. PMID 23691202
- [Background] Corso A, Lorenzi A, Terulla V, Airo F, Varettoni M, Mangiacavalli S, Zappasodi P, Rusconi C, Lazzarino M. Modification of thrombomodulin plasma levels in refractory myeloma patients during treatment with thalidomide and dexamethasone. Ann Hematol. 2004 Sep;83(9):588-91. doi: 10.1007/s00277-004-0891-6. Epub 2004 Jul 3. PMID 15235749
- [Background] Pal R, Monaghan SA, Hassett AC, Mapara MY, Schafer P, Roodman GD, Ragni MV, Moscinski L, List A, Lentzsch S. Immunomodulatory derivatives induce PU.1 down-regulation, myeloid maturation arrest, and neutropenia. Blood. 2010 Jan 21;115(3):605-14. doi: 10.1182/blood-2009-05-221077. Epub 2009 Nov 25. PMID 19965623
- [Background] Palumbo A, Cavo M, Bringhen S, Zamagni E, Romano A, Patriarca F, Rossi D, Gentilini F, Crippa C, Galli M, Nozzoli C, Ria R, Marasca R, Montefusco V, Baldini L, Elice F, Callea V, Pulini S, Carella AM, Zambello R, Benevolo G, Magarotto V, Tacchetti P, Pescosta N, Cellini C, Polloni C, Evangelista A, Caravita T, Morabito F, Offidani M, Tosi P, Boccadoro M. Aspirin, warfarin, or enoxaparin thromboprophylaxis in patients with multiple myeloma treated with thalidomide: a phase III, open-label, randomized trial. J Clin Oncol. 2011 Mar 10;29(8):986-93. doi: 10.1200/JCO.2010.31.6844. Epub 2011 Jan 31. PMID 21282540
- [Background] Larocca A, Cavallo F, Bringhen S, Di Raimondo F, Falanga A, Evangelista A, Cavalli M, Stanevsky A, Corradini P, Pezzatti S, Patriarca F, Cavo M, Peccatori J, Catalano L, Carella AM, Cafro AM, Siniscalchi A, Crippa C, Petrucci MT, Yehuda DB, Beggiato E, Di Toritto TC, Boccadoro M, Nagler A, Palumbo A. Aspirin or enoxaparin thromboprophylaxis for patients with newly diagnosed multiple myeloma treated with lenalidomide. Blood. 2012 Jan 26;119(4):933-9; quiz 1093. doi: 10.1182/blood-2011-03-344333. Epub 2011 Aug 11. PMID 21835953
- [Background] Chakraborty R, Bin Riaz I, Malik SU, Marneni N, Mejia Garcia A, Anwer F, Khorana AA, Rajkumar SV, Kumar S, Murad MH, Wang Z, Khan SU, Majhail NS. Venous thromboembolism risk with contemporary lenalidomide-based regimens despite thromboprophylaxis in multiple myeloma: A systematic review and meta-analysis. Cancer. 2020 Apr 15;126(8):1640-1650. doi: 10.1002/cncr.32682. Epub 2020 Jan 8. PMID 31913498
- [Background] de Waal E. Multiple aspects of a plasma cell dyscrasia [PhD]. University of Groningen; 2018